CLINICAL TRIAL: NCT02819050
Title: A Prospective Randomized Controlled Tiral Comparing Sprinting Versus Non-sprinting Approach to Wean Nasal Continous Positive Airway Pressure Support in Premature Infants Born at Less Than 30 Weeks Gestational Age
Brief Title: Effective Approaches & Strategies to Ease Off Nasal CPAP In Preterm Infants
Acronym: EASEOFFNCPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Virender Rehan, MD, Chair, Department of Neonatology, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30166-01
Record Dates: First submitted 2016-05-24; First posted 2016-06-30 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Neonatal Respiratory Distress Syndrome; Extremely Low Birth Weight Infant (ELBW); BronchoPulmonary Dysplasia
Keywords: CPAP; Extremely Low Birth Weight Infant (ELBW); Non-invasive respiratory support; Premature infants; Non invasive ventilation weaning
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sprinting (Experimental): Take off NCPAP twice daily for 3hours (day 1), Take off NCPAP twice daily for 6hours (day 2), Take off NCPAP twice daily for 9hours (day 3), Placed back on NCPAP for 24hours (day 4), Switch to nasal cannula at a flow rate of 1.5-2 L/min (day 5)
  Interventions: Device: NCPAP
- Non-Sprinting (Active Comparator): * If the infant was on NCPAP 6, Infant was weaned down to CPAP 5 for 96 hours. If they met stability criteria, then infant was switched to room air (no flow) or no more than 2L NC.
  * If the infant was on NCPAP 5, the infant was continued on CPAP 5 for 96 hours If they met stability criteria, then infant was switched to room air (no flow) or no more than 2L NC.
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: NCPAP — Nasal Continuous Positive Airway Pressure

SUMMARY:
Though Nasal Continuous Positive Airway Pressure (NCPAP) is a commonly used form of non-invasive neonatal respiratory support, the optimal method of weaning off NCPAP is not well established. In this prospective, two-center randomized control trial we hypothesize that gradually increasing time off NCPAP (sprinting) increases the success of weaning NCPAP off in infants born between 23 0/7-30 6/7 weeks of gestational age.

DETAILED DESCRIPTION:
Eligible infants admitted to two Neonatal Intensive Care Units (NICUs) were randomized to a sprinting (SP) vs. a non-sprinting (NSP) protocol, both over 4 days. Infants assigned to the SP group sprinted twice daily for 3h (day 1), 6h (day 2), 9h (day 3) & then 24h back on NCPAP (day 4) before switching to nasal cannula (NC) on day 5. Infants in the NSP group were maintained on NCPAP of 5 cm of water for the first 4 days before switching to NC on day 5, similar to the SP group. Infants in both groups were observed for the next 3 days (day 5-7) to ensure stability off CPAP

ELIGIBILITY:
Inclusion Criteria:

* Born between 23 0/7 - 30 6/7 weeks GA
* At least 26 0/7 weeks corrected GA.
* On NCPAP for at least 24 hours
* Stable on ≤0.3 FiO2 for at least 24 hours

Initiation of study protocol, i.e., weaning from NCPAP, was started when infant met all of the following criteria for at least 24 hours:

* Requiring NCPAP of 4-6 cm of H2O and FiO2 ≤0.3.
* All babies < 32 weeks corrected GA should have been loaded or already on maintenance caffeine (caffeine citrate 20 mg/kg as the loading and 5-10 mg/kg as the maintenance dose).
* Stable respiratory system assessment (respiratory rate of < 70/min, no significant chest retractions (sternal/ diaphragmatic), and baseline oxygen saturation > 86%) and otherwise deemed clinically stable for weaning off non-invasive ventilation by medical team
* If post-surgery, infant must be at least 2 weeks post-operative and off antibiotics with no concern or need for repeat surgery.
* A documented hemoglobin of more than 8 g/dl within 7 days of initiation of the study.
* Meeting "stability criteria" defined below:

  * The infant had to be tolerating a flow of no more than 2 liters NC on a FiO2 of 0.30 or less to keep oxygen saturations above 85% (should match what you wrote below in failure criteria)%.
  * Have a respiratory rate of less than 70 on average over 24 hours for more than 24 hours
  * The infant could have no significant chest recession (sternal/diaphragmatic)

Exclusion Criteria:

* Evidence of a hemodynamically or clinically significant (worsening respiratory status or pulmonary edema on chest x-ray) Patent ductus arteriosus, diagnosed either clinically or echocardiographically.

  * Any significant congenital abnormality (abnormalities affecting a major organ system, airway, or musculoskeletal system).
  * Hemodynamic/respiratory instability or currently being treated for suspected or proven sepsis (positive blood culture)
  * Grade IV intraventricular hemorrhage
  * Inability to obtain informed parental consent

Min Age: 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virender Rehan, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Finer NN, Carlo WA, Duara S, Fanaroff AA, Donovan EF, Wright LL, Kandefer S, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Delivery room continuous positive airway pressure/positive end-expiratory pressure in extremely low birth weight infants: a feasibility trial. Pediatrics. 2004 Sep;114(3):651-7. doi: 10.1542/peds.2004-0394. PMID 15342835
- [Background] Vaucher YE, Peralta-Carcelen M, Finer NN, Carlo WA, Gantz MG, Walsh MC, Laptook AR, Yoder BA, Faix RG, Das A, Schibler K, Rich W, Newman NS, Vohr BR, Yolton K, Heyne RJ, Wilson-Costello DE, Evans PW, Goldstein RF, Acarregui MJ, Adams-Chapman I, Pappas A, Hintz SR, Poindexter B, Dusick AM, McGowan EC, Ehrenkranz RA, Bodnar A, Bauer CR, Fuller J, O'Shea TM, Myers GJ, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network. Neurodevelopmental outcomes in the early CPAP and pulse oximetry trial. N Engl J Med. 2012 Dec 27;367(26):2495-504. doi: 10.1056/NEJMoa1208506. PMID 23268664
- [Background] Singh SD, Bowe L, Clarke P, Glover K, Pasquill A R, MJ et al. Is decreasing pressure or increasing time off the better strategy in weaning VLBW infants from nasal CPAP? Eur J Pediatr B Abstr Eur Acad Pediatr. 2006;Abstract.
- [Background] A Soe, J Hodgkinson, B Jani DAD. Nasal continous positive airway pressure weaning in preterm infants. Eur J Pediatr B Abstr Eur Acad Pediatr. 2006;Abstract.
- [Background] Todd DA, Wright A, Broom M, Chauhan M, Meskell S, Cameron C, Perdomi AM, Rochefort M, Jardine L, Stewart A, Shadbolt B. Methods of weaning preterm babies <30 weeks gestation off CPAP: a multicentre randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F236-40. doi: 10.1136/adc.2011-300133. Epub 2012 May 18. PMID 22611116
- [Background] Jardine LA, Inglis GD, Davies MW. Strategies for the withdrawal of nasal continuous positive airway pressure (NCPAP) in preterm infants. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD006979. doi: 10.1002/14651858.CD006979.pub2. PMID 21328289
- [Background] Rastogi S, Rajasekhar H, Gupta A, Bhutada A, Rastogi D, Wung JT. Factors Affecting the Weaning from Nasal CPAP in Preterm Neonates. Int J Pediatr. 2012;2012:416073. doi: 10.1155/2012/416073. Epub 2011 Dec 8. PMID 22187570
- [Background] Rastogi S, Wong W, Gupta A, Bhutada A; Deepa Rastogi; Maimonides Neonatal Group. Gradual versus sudden weaning from nasal CPAP in preterm infants: a pilot randomized controlled trial. Respir Care. 2013 Mar;58(3):511-6. doi: 10.4187/respcare.01999. PMID 22906960
- [Derived] Eze N, Murphy D, Dhar V, Rehan VK. Comparison of sprinting vs non-sprinting to wean nasal continuous positive airway pressure off in very preterm infants. J Perinatol. 2018 Feb;38(2):164-168. doi: 10.1038/jp.2017.161. Epub 2017 Oct 26. PMID 29072676

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Sprinting: * If the infant was on NCPAP 6, Infant was weaned down to CPAP 5 for 96 hours. If they met stability criteria, then infant was switched to room air (no flow) or no more than 2L NC.
  * If the infant was on NCPAP 5, the infant was continued on CPAP 5 for 96 hours If they met stability criteria, then infant was switched to room air (no flow) or no more than 2L NC.
  NCPAP: Nasal Continuous Positive Airway Pressure
Period: Overall Study
Arm/Group | Sprinting | Non-Sprinting
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sprinting | Non-Sprinting | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: Weeks] | 33.4 [28.7 to 41.4] | 33.2 [29.9 to 36.6] | 33.3 [28.7 to 41.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 19 | 15 | 34
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Wean Off CPAP at the First Attempt
Description: Measured by successful wean off CPAP on first attempt, i.e., no NCPAP requirement after 7 days on wean protocol on first attempt.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sprinting | Non-Sprinting
Number analyzed (Participants) | 40 | 40
Participants | 31 | 30

2. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia
Description: Measured as an oxygen requirement at 36 weeks corrected gestational age
Time Frame: 1-2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sprinting | Non-Sprinting
Number analyzed (Participants) | 40 | 40
Participants | 11 | 14

3. Secondary Outcome: Number of Participants With Retinopathy of Prematurity (ROP)
Description: Measured as clinical signs of stage 2 or above ROP on retinal exam prior to discharge
Time Frame: 1-2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Sprinting | Sprinting
Number analyzed (Participants) | 40 | 40
Participants | 12 | 15

4. Secondary Outcome: Number of Participants With Periventricular Leukomalacia (PVL)
Description: Measured as radiologic findings of PVL noted prior to discharge
Time Frame: 1-2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sprinting | Non-Sprinting
Number analyzed (Participants) | 40 | 40
Participants | 0 | 1

5. Secondary Outcome: Length of Stay (Days)
Description: Measures as the number of days patient remained hospitalized after birth at the study hospital.
Time Frame: 60-108 days
Measure: Median (Full Range); unit: Days
Arm/Group | Non-Sprinting | Sprinting
Number analyzed (Participants) | 40 | 40
Days | 82.5 [60.5 to 103.3] | 78 [62 to 108]

6. Secondary Outcome: Corrected Gestational Age at Time of Discharge/Transfer
Description: Measured as the corrected gestational age at which the patient was discharged or transferred.
Time Frame: 36weeks-41weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Non-Sprinting | Sprinting
Number analyzed (Participants) | 40 | 40
weeks | 33.4 [28.7 to 41.4] | 33.2 [29.9 to 36.6]

7. Secondary Outcome: Number of Attempts to Wean Off CPAP
Description: Number of attempts made to wean off CPAP
Time Frame: Until completely weaned off CPAP
Measure: Median (Full Range); unit: Attempt
Arm/Group | Non-Sprinting | Sprinting
Number analyzed (Participants) | 40 | 40
Attempt | 1 [1 to 2] | 1 [1 to 2]

8. Secondary Outcome: Number of Days on Protocol
Description: Measured as the total number of days the patient was on the study protocol
Time Frame: 7-10 days
Measure: Median (Full Range); unit: Days
Arm/Group | Non-Sprinting | Sprinting
Number analyzed (Participants) | 40 | 40
Days | 7 [7 to 7] | 7 [7 to 10]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Sprinting | Non-Sprinting
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
Limitations:

1. A non-blinded study.
2. Relative imbalance in the number of infants included at the two study sites
3. Inadequate sample size for data analysis based on GA sub-stratification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No